CLINICAL TRIAL: NCT03147092
Title: Matão Controlling Hypertension (MatCH Study): Rationale and Design. Project to Reduce Incidence of Arterial Hypertension in City of Matão, Brazil.
Brief Title: Matão Controlling Hypertension (MatCH Study): Rationale and Design
Acronym: MatCH
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Neurológico de Pesquisa e Reabiitação, Brazil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMinelli
Record Dates: First submitted 2017-04-30; First posted 2017-05-10 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-04

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Captopril; Hydrochlorothiazide; Tablets; Atenolol; Losartan; Clonidine

STUDY DESIGN:
Intervention Model Description: A single group of hypertensive individuals will be submitted to same treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertension group (Experimental): Hypertensive patients will be counseled to initiate life style changes as weight loss, salt reduction, exercise, reduced alcohol consumption, smoking cessation and fresh fruits and vegetables in their diets. Drug treatment will be started for subjects that are not responding to nonpharmacological treatment. The anti-hypertensive medications will be Captopril 25Mg, Hydrochlorothiazide 25Mg Oral Tablet, atenolol and Losartan potassium 50 mg. All of these anti-hypertensive drugs are available in the PPP. If BP control is not yet obtained, other antihypertensive drugs will be requested: clonidine, spironolactone, hydralazine and amlodipine.
  Interventions: Drug: Captopril 25Mg, Hydrochlorothiazide 25Mg Oral Tablet,; Drug: Atenolol; Drug: Losartan potassium 50mg; Drug: Clonidine

INTERVENTIONS:
Drug: Captopril 25Mg, Hydrochlorothiazide 25Mg Oral Tablet, — Treatment of hypertensive subjects
Drug: Atenolol — Treatment of hypertensive subjects
Drug: Losartan potassium 50mg — Treatment of hypertensive subjects
Drug: Clonidine — Treatment of hypertensive subjects

SUMMARY:
Background Hypertension is the main risk factor for most cardiovascular diseases. Blood pressure (BP) control has been shown to reduce the incidence of stroke, myocardial infarction, renal diseases and heart failure. Although BP lowering is effective, few population programs can achieve BP control. A coordinated and organized system from the Brazilian Ministry of Healthy involving Family Health Strategy (FHS), a program for the prevention of chronic disease, and the Popular Pharmacy Program (PPP), which subsidizes medications for the population, could allow an earlier identification and better BP control. Matão Controlling Hypertension (MatCH) is a community-based population project that aims to apply an organized, integrated and coordinated program in the city of Matão, Brazil, involving FSH and PPP in order to actively search, treat and follow-up hypertensive subjects.

Method This is a population community-based, prospective, interventional, follow-up study where all subjects aged ≥ 40 years assisted by the FHS program in Matão will have BP assessed monthly by trained Community Health Agents (CHA) during a domiciliary visit. Identified hypertensive subjects will be referred to FHS physicians for nonpharmacological and pharmacological treatment. Most of the hypertensive drugs used will be available thought the PPP. Prevalence of hypertension, awareness, demographics and risk factors will be correlated with BP control. The population study is expected to involve approximately 15,000 subjects. The study period will be four years.

Discussion Considering that hypertension is asymptomatic in most cases, to reduce the population burden of BP-related deaths and diseases it is essential to detect and treat early all hypertensive patients. If BP control be achieved on a large scale, this program can be applied to other populations from developing countries.

DETAILED DESCRIPTION:
Hypertension is the main risk factor associated with the global burden of disease and mortality.

Brazil, a middle-income country and the largest in Latin America, has a prevalence of hypertension of about 35% (Ribeiro AL et al, 2016), with no significant difference between genders.

A decrease in cardiovascular disease mortality has been observed. This phenomenon could be attributed to some public healthy preventive programs such as the Family Healthy Strategy (FHS) (Macinko J et al, 2015) and the Popular Pharmacy Program (PPP) (Emmerick I et al, 2015), both supported by the Brazilian Ministry of Healthy. FHS is focused on a community-based approach to providing primary health care. Physicians, nurses, and community health agents (CHA) visit residents in their homes to prevent complications and to take care of chronic diseases.

The purpose of the Matão Controlling Hypertension (MatCH) project is to apply an organized, integrated and coordinated program of all health services in Matão, mainly involving FSH and PPP, for an earlier identification of hypertensive individuals, followed by treatment and follow-up in order to control their BP.

Objective

1. To identify hypertensive subjects aged ≥ 40 years in a defined population.
2. To control BP in this population by the optimization of the local public health system.

   Hypothesis

   A better BP control can be obtained with an integrated and coordinated hypertension detection and control system involving the Family Healthy Strategy (FHS), Popular Pharmacy Program (FPP) and local public health services in a defined Brazilian population.

   Methods

   Study design

   This will be a population-based, prospective, interventional, follow-up study.

   Inclusion criteria All consented subjects aged ≥ 40 years belonging to FHS and residing in Matão.

   Exclusion criteria Patients younger than 40 years. Subjects not belonging to FHS in Matão. Subjects from other cities.

   Study period Four years

   Outcomes

   Primary outcomes Prevalence of hypertension at initial assessment. Number of hypertensive subjects with BP controlled during follow-up .

   Secondary outcomes

   Correlation of hypertension prevalence and BP control with demographics, risk factors and end organ diseases.

   Baseline procedures

   Matão city characteristics

   The study will be conducted in Matão, Brazil, a city located in São Paulo state, the wealthiest state in Brazil, in the Brazilian southwest, 300 km northwest to the state capital. According to the 2010 Brazilian census, the Matão population was 76,786 and the estimate for 2017 was 81,878 inhabitants, with no difference in sex distribution . The economy is mainly based on industrial activities and on general services. Ethnicity is diverse, but most people are of Caucasian origin, descendants of European immigrants. The population is urban and stable, with a low rate of interurban migration. About 95% of all dwellings have piped water, a sewage network and electricity.

   The public healthy system of Matão is well organized. As is the case for most Brazilian cities, Matão has FHS. There are 12 FHS in the city covering a population of 44,850 people, representing about 57% of the whole population. The city also participates in the PPP.

   Study population The 2010 Brazilian census indicated that 29,192 Matão inhabitants were ≥ 40 years old, representing 38% of the total population. Considering a population of 41,400 covered by FHS, 38% of >40-year-old subjects represent a study population of about 15,000 subjects. The reason to include a population aged ≥ 40 years is justified by the fact that the prevalence of hypertension is almost 20% among subjects 35 to 44 years of age.

   BP assessment BP will be measured by the CHA using the automated device Omron M2® validated. The CHA will be trained to measure BP properly according to the following protocol (Malachias et al, 2016): BP will be measured in both arms; if the readings are different, the arm with the higher reading will be used for subsequent measurements made 1 to 2 minutes apart and the average of these measurements will be considered. A wider cuff will be used for patients with an arm circumference of more than 32 cm.

   Definitions and classifications

   Hypertension diagnosis

   The diagnosis of hypertension will be confirmed if systolic blood pressure is ≥ 140 mmHg or diastolic pressure is ≥ 90 mmHg, or both, in two different measurements separated by about 30 days (Malachias M et al, 2016).

   Controlled BP will be defined as systolic blood pressure ≤ 139 mmHg and diastolic blood pressure ≤ 89 mmHg.

   Follow-up

   The BP of the study population will be measured monthly by CHA. If BP is above normal ranges and continues to be elevated at the second monthly measurement, the subject will be followed up more closely by the FHS physician, who will decide the best hypertensive treatment strategy. If BP continues to be elevated at the monthly assessments, even with optimized treatment, the subject will be referred to and followed up by the cardiologist from the public health service connected to FHS. The monthly BP values obtained will be inserted in a data base and software developed by the research team.

   Subject evaluation

   Questionnaire

   Subject data will be collected with a structured questionnaire about age, gender, years of education, previous history of hypertension, stroke, coronary artery disease, chronic kidney disease, diabetes mellitus, peripheral artery disease, dyslipidemia, alcohol abuse, smoking, and physical activity.

   Treatment of hypertension

   The treatment of hypertension will be based on the recent VII Brazilian Guidelines of Arterial Hypertension. (Malaquias M et al, 2016)

   Nonpharmacological treatment All hypertensive patients will be counseled to initiate life style changes. They will receive verbal and written orientations regarding weight loss, salt reduction, exercise, reduced alcohol consumption, smoking cessation, and the introduction of more fresh fruits and vegetables in their diets.

   Pharmacological treatment

   Drug treatment will be started for subjects with BP ≥140/90 mm Hg at second assessment, those with SBP≥ 180 mmHg and/or DBP ≥ 110 mmHg at first assessment and all hypertensive subjects that are not responding to nonpharmacological treatment.

   In a first step, the first lines of anti-hypertensive medication will be the angiotensin-converting enzyme inhibitors (ACEI) captopril and enalapril, or the angiotensin receptor blocker (ARB) losartan, or calcium channel blockers (CCB), nifedipine, diltiazem and verapamil, or diuretics, the thiazide-type diuretic hydrochlorthiazide or chlortalidone, or beta-blockers, atenolol, in selected cases. In a second step, if BP is not controlled, a combination of two drug classes will be tried. If BP is not achieved, in a third step, a third drug class will be added. All of these anti-hypertensive drugs are available in the PPP. In a fourth step, when BP control is not yet obtained, other antihypertensive drugs will be requested from the city public health department, preferably low costs drugs such as clonidine, spironolactone, hydralazine and amlodipine. During this phase, a consultation with a hypertension specialist physician will be provided. The combined use of ACEI and ARB will be avoided. For individuals with chronic kidney disease, initial antihypertensive treatment will include an ACEI or ARB. This includes all chronic kidney disease patients with hypertension independent of diabetes and race.

   Ethical approval

   The project was approved by the Ethics Committee of Universidade de Araraquara, which is accredited by the Office of Human Research Protections as an Institutional Review Board, process no 1.985.885. All participants will give written informed consent to participate.

   Statistical analysis

   To analyze the associations between the prevalence of hypertension at baseline, demographic variables, risk factors and end organ diseases the Chi-square test will be used for categorical variables and one-way ANOVA for numeric variables. Logistic regression will be used for multivariate analysis. Since BP will be assessed monthly, the mean BP values for each month will be compared by ANOVA for multiple repeated measurements. After the second assessment at baseline to determine how many hypertensive subjects achieved BP control, the McNemar test for paired samples will be used. For all tests, will be considered a level of significance of 5% and a 95% confidence interval (CI).

   Discussion

   Hypertension control on a large scale can be a challenge, with barriers attributed to patients, healthcare providers, health-care systems, and the silent nature of the disease (Arima H et al 2011).

   Community resources such as volunteers, health nurses, and local organizations are underutilized to support disease prevention and primary health care. Synergy created by connecting family physicians, patients, peer volunteers and local resources can lead to better health outcomes for community residents (Ye et al, 2013).

   The purpose of this present study is in accordance with these studies. The differential is that it will be applied to a larger population through local health services with the efforts involving the CHA from the FHS program. This model of BP control will be tested in a community-based population, i.e., in the real world, and not in a selected sample that could generate undesirable bias analysis.

   The project has many positive aspects. The local health care system has already been structured. No additional cost will be necessary regarding human resources or new buildings and most of the antihypertensive drugs are available at PPP. Individuals aged ≥ 40 years will be included, so that it will be possible to identify and reduce earlier the risk of cardiovascular disease in hypertensive patients.

   The possible disadvantage would be the high cost to reach a large population. However, the financial resources of FHS are the same as those already implemented for five years. Not all recommended anti-hypertensive drugs will be immediately available for pharmacological treatment.

   Some challenges are expected. In a pilot study (Minelli et al, 2016), almost 50% of cases was not possible to assess BP during CHA visits. Most of the subjects were out working and a minority refused to take BP assessment. An alternative to this problem is to make an appointment with these missing subjects or to visit them at their local jobs. Another challenge is to convince the target population to take their medications even if there are no hypertension-related symptoms.

   This project is a proof of concept, i.e., it shows that it is feasible to control BP at levels better than the reported 40% BP control among Brazilian hypertensive subjects, in a large number of people, using a system that already exists, i.e., FHS, PPP and local public health services, although with a coordinated, centralized and organized program directed at BP control.

   If the goals of large-scale BP control be achieved, this model can be applied to other vulnerable populations from developing countries.

ELIGIBILITY:
Inclusion Criteria:

* All consented subjects aged ≥ 40 years belonging to Family Strategy Health program and residing in Matão.

Exclusion Criteria:

* Patients younger than 40 years.
* Subjects not belonging to Family Strategy Health program in Matão.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of hypertensive subjects with BP controlled during follow-up | Through study completion, an average of 2 years
  Controlled BP will be defined as systolic blood pressure ≤ 139 mmHg and diastolic blood pressure ≤ 89 mmHg.

SECONDARY OUTCOMES:
Correlation of BP control with demographics | Through study completion, an average of 3 years
  Age, gender, years of education.
Correlation of BP control with risk factors | Through study completion, an average of 3 years
  Previous history of hypertension, diabetes mellitus, dyslipidemia, alcohol abuse, smoking, and physical activity
Correlation of BP end organ disease | Through study completion, an average of 3 years.
  previous history of stroke, coronary artery disease, chronic kidney disease, peripheral artery disease.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Minelli, MD, PhD, Principal Investigator — Hospital Carlos Fernando Malzoni

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ribeiro AL, Duncan BB, Brant LC, Lotufo PA, Mill JG, Barreto SM. Cardiovascular Health in Brazil: Trends and Perspectives. Circulation. 2016 Jan 26;133(4):422-33. doi: 10.1161/CIRCULATIONAHA.114.008727. PMID 26811272
- [Result] Macinko J, Harris MJ. Brazil's family health strategy--delivering community-based primary care in a universal health system. N Engl J Med. 2015 Jun 4;372(23):2177-81. doi: 10.1056/NEJMp1501140. No abstract available. PMID 26039598
- [Result] Emmerick IC, do Nascimento JM Jr, Pereira MA, Luiza VL, Ross-Degnan D; ISAUM-Br Collaborative Group. Farmacia Popular Program: changes in geographic accessibility of medicines during ten years of a medicine subsidy policy in Brazil. J Pharm Policy Pract. 2015 Mar 9;8(1):10. doi: 10.1186/s40545-015-0030-x. eCollection 2015. PMID 25926990
- [Result] Malachias MVB, Gomes MAM, Nobre F, Alessi A, Feitosa AD, Coelho EB. 7th Brazilian Guideline of Arterial Hypertension: Chapter 2 - Diagnosis and Classification. Arq Bras Cardiol. 2016 Sep;107(3 Suppl 3):7-13. doi: 10.5935/abc.20160152. No abstract available. PMID 27819381
- [Result] Malachias MVB, Paulo Cesar Veiga Jardim PCV Junior, Almeida FA, Lima E Junior, Feitosa GS. 7th Brazilian Guideline of Arterial Hypertension: Chapter 7 - Pharmacological Treatment. Arq Bras Cardiol. 2016 Sep;107(3 Suppl 3):35-43. doi: 10.5935/abc.20160157. No abstract available. PMID 27819386
- [Result] Arima H, Barzi F, Chalmers J. Mortality patterns in hypertension. J Hypertens. 2011 Dec;29 Suppl 1:S3-7. doi: 10.1097/01.hjh.0000410246.59221.b1. PMID 22157565
- [Result] Minelli C, Borin LA, Trovo Mde C, Dos Reis GC. Hypertension Prevalence, Awareness and Blood Pressure Control in Matao, Brazil: A Pilot Study in Partnership With the Brazilian Family Health Strategy Program. J Clin Med Res. 2016 Jul;8(7):524-30. doi: 10.14740/jocmr2582w. Epub 2016 May 29. PMID 27298661
- See also: Family Health Strategy Program, extension — http://dab.saude.gov.br/portaldab/historico_cobertura_sf.php/UnidadeGeográfica/SãoPaulo/Matão/Período2016